CLINICAL TRIAL: NCT01286051
Title: Efficacy of Single Dose Ganirelix in Gonadotropin Ovulation Induction Cycles
Brief Title: Single Injection of Ganirelix in Gonadotropin Intrauterine Insemination (IUI) Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Houston Fertility Institute (Other)
Responsible Party: Principal Investigator, Ghassan F. Haddad, Medical Director, Houston Fertility Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P08115
Record Dates: First submitted 2011-01-25; First posted 2011-01-31 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Compare Pregnancy Rates Between FSH Stimulation and FSH and; GnRH Antagonist
Keywords: ovulation induction, GnRH
MeSH Terms: interventions — follitropin beta; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follistim (Active Comparator): standard treatment
  Interventions: Drug: Follistim administration
- Follistim plus single ganirelix injection (Experimental)
  Interventions: Drug: Follistim plus Ganirelix

INTERVENTIONS:
Drug: Follistim administration — adminstation of FSH for ovulation induction
  Other Names: Follistim
  Arms: Follistim
Drug: Follistim plus Ganirelix — Follistim plus single injection of ganirelix
  Other Names: Follistim; ganirelix
  Arms: Follistim plus single ganirelix injection

SUMMARY:
Ovulation induction (OI) using gonadotropins is one of the most widely prescribed treatments of infertility. One common problem encountered while attempting OI using gonadotropins is premature ovulation. The purpose of this study is to examine the effect of a single injection of a medication, called ganirelix, to prevent premature ovulation. Patients will be divided into two groups. In the first group, gonadotropins will be used to stimulate the ovaries. In the second group gonadotropins will be used in addition to a single injection of ganirelix, a gonadotropin releasing hormone (GnRH) antagonist. Pregnancy rates will be compared between groups.

DETAILED DESCRIPTION:
A randomized prospective study will be performed on patients attempting pregnancy using ovulation induction/intra-uterine insemination (IUI). Patients will be randomly assigned to one of two protocols:

Protocol A (control group): On menstrual cycle day 3, the patient will start gonadotropins (Follistim) injections at a starting dose of 75-150 IU and monitored according to the discretion of the treating physician. When the leading follicle reaches a size of at least 18mm, intramuscular human chorionic gonadotripin (hCG) (10,000 IU) is administered, followed by two inseminations, one at 12 hours after hCG, and the other at 36 hours. All patients will have luteal support using progesterone vaginal suppositories at a dose of 200mg two times per day (BID). Pregnancy testing will be scheduled at 2 weeks after the IUI. The treatment cycle typically lasts from 8-13 days, depending on the patient's response.

Protocol B (study group): On menstrual cycle day 3, the patient will start gonadotropins (Follistim) injections at a starting dose of 75-150 IU and monitored according to the discretion of the treating physician. When the leading follicle reaches a size of 13-14mm in mean diameter, or when the estradiol level reaches a level of 400 pg/ml, ganirelix injection at the standard dose of 250mcg is given once subcutaneously. When the leading follicle reaches a size of at least 18mm, intramuscular hCG (10,000IU) is administered followed by two inseminations, one at 12 hours after hCG, and the other at 36 hours. All patients will have luteal support using progesterone suppositories at a dose of 200mg BID. Pregnancy testing will be scheduled at 2 weeks after the IUI. The treatment cycle typically lasts from 8-13 days, depending on the patient's response.

Patients will be randomized, via computer generated program, in a 1:1 fashion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ovulation induction (OI) between ages 18 - 39 years.
* One or more of the following infertility diagnoses: ovulation dysfunction, mild male factor infertility (sperm concentration of 5- 20 million/ml, and/or sperm motility 10% - 40%) , absence teratospermia (i.e. strict morphology > 4%), unexplained infertility.
* Patent Fallopian tubes.
* Normal uterine structure (i.e. absence of mullerian anomalies)
* Ability to consent to the study.
* Patients should be Houston Fertility Institute patients

Exclusion Criteria:

Exclusion criteria include:

* Age 39 or above
* Severe male factor (concentration < 10 million/ml or strict morphology < 4%)
* Obstructed Fallopian tubes on one or both sides
* Stage III or IV endometriosis
* Elevated FSH level (>10 IU/L)
* Low antral follicular count (< 4 antral follicles per ovary)
* Any other contraindication for ovulation induction
* Inability to consent to the study
* History of any prior failed OI/IUI cycle

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pregnancy rates | One cycle of controlled ovarian stimulation (one month)
  Follicle stimulating hormone (FSH) and IUI

SECONDARY OUTCOMES:
Premature leuteinizing hormone (LH) surge and ovulation | One cycle of controlled ovarian stimulation (one month)
  pregnancy rate in one cycle of FSH and single injection of GnRH antagonist

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan F Haddad, M.D., Principal Investigator — Houston Fertility Institute
Locations (1):
- Houston Fertility Institute, Houston, Texas, United States

REFERENCES:
- See also: practice website — http://www.hfi-ivf.com